CLINICAL TRIAL: NCT00539760
Title: A Phase I, Randomized, Observer- and Subject-Blind, Placebo-Controlled, Single Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK1827771 in Healthy Volunteers
Brief Title: A Phase I Rheumatoid Arthritis Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 110394
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Arthritis, Rheumatoid
Keywords: domain antibody; Rheumatoid Arthritis,
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Subjects receiving GSK 1827771 in sub-cohort Xa (Cohort 1-5) (Experimental): Eligible subjects will receive GSK1827771 with the starting dose of 0.3 milligram (mg)
  Interventions: Drug: GSK1827771
- Subjects receiving placebo in sub-cohort Xa (Cohort 1-5) (Placebo Comparator): Eligible subjects will receive placebo matching to GSK1827771
  Interventions: Drug: Placebo
- Subjects receiving GSK 1827771 in sub-cohort Xb (Cohort 1-5) (Experimental): Eligible subjects will receive GSK1827771 via injection
  Interventions: Drug: GSK1827771
- Subjects receiving placebo in sub-cohort Xb (Cohort 1-5) (Placebo Comparator): Eligible subjects will receive placebo matching to GSK1827771
  Interventions: Drug: Placebo
- Subjects receiving GSK 1827771 in sub-cohort Xc (Cohort 1-5) (Experimental): Eligible subjects will receive GSK1827771 via injection
  Interventions: Drug: GSK1827771
- Subjects receiving placebo in sub-cohort Xc (Cohort 1-5) (Placebo Comparator): Eligible subjects will receive placebo matching to GSK1827771
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1827771 — GSK1827771 will be administered using injection via subcutaneous (SC) route.
  Arms: Subjects receiving GSK 1827771 in sub-cohort Xa (Cohort 1-5); Subjects receiving GSK 1827771 in sub-cohort Xb (Cohort 1-5); Subjects receiving GSK 1827771 in sub-cohort Xc (Cohort 1-5)
Drug: Placebo — Placebo to GSK1827771 for Injection will be administered via SC route
  Arms: Subjects receiving placebo in sub-cohort Xa (Cohort 1-5); Subjects receiving placebo in sub-cohort Xb (Cohort 1-5); Subjects receiving placebo in sub-cohort Xc (Cohort 1-5)

SUMMARY:
GSK182771 is a domain antibody targeting the interleukin (IL)-1 receptor which is being developed for the treatment of rheumatoid arthritis. This study is being done in healthy volunteers to verify the safety and tolerability of GSK182771

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men or women as determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests and cardiac assessment.
* Female subjects of non-childbearing potential.
* Male subjects must agree to abstain from or agree to use adequate contraception, in addition to having their female partner use another form of contraception. This criterion must be followed from the time of the first dose of study medication until Pharmacokinetic levels are determined to be below the LLQ.
* Men or women who are between 18 and 55 years of age, inclusive.
* Body Mass Index (BMI) within the range of 18-35 kilogram per meter square (kg/m^2) inclusive.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* The subject has a positive pre-study urine drug/urine alcohol screen. A minimum list of drugs that will be screened for includes amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A history of regular alcohol consumption averaging >7 drinks/week for females or >14 drinks/week for males. One drink is equivalent to (12 g alcohol) = 5 ounces [150 milliliter (mL)] of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits
* The subject is unwilling to abstain from alcohol consumption from 48 hour prior to dosing until discharge from the clinic, and for 48 hour prior to all other out-patient clinic visits.
* Smoked or used tobacco or nicotine-containing products within the previous 6 months prior to the first dose of current study medication.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Previous exposure to or treatment with PEGylated molecules.
* Use of anti-Tumor Necrosis Factor (anti-TNF) drugs within 60 days prior to dosing.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days , or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy (including antibiotics) which, in the opinion of the investigator and/or GSK Medical Monitor, contraindicates the subject's participation.
* Positive pregnancy test at Screening or on Day -1 (females only).
* Any clinically significant abnormality identified on the screening medical assessment or examination, or ECG.
* Any white blood cell (WBC) or neutrophil count outside the normal range at screening or on Day -1.
* History of significant cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal conditions that in the opinion of the investigator and/or GSK Medical Monitor, places the subject at an unacceptable risk as participant in this trial.
* History of any autoimmune or current inflammatory conditions including rheumatoid arthritis or any other joint disease.
* History of malignancy, except for surgically cured basal cell carcinoma or cured cervical carcinoma (> 2 yrs prior to dosing).
* Currently has asthma or history of chronic obstructive pulmonary disease (COPD).
* Current evidence of ongoing or acute infection.
* The subject has a history of repeated, chronic or opportunistic infections which, in the opinion of the investigator and/or GSK Medical Monitor, places the subject at an unacceptable risk as a participant in this trial.
* History of Mycobacterium tuberculosis or any other previous Mycobacterium infection.
* A positive pre-study Hepatitis B surface antigen, positive Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody testing result.
* History of a severe allergic reaction, angio-edema, anaphylaxis or immunodeficiency
* History of elevated blood pressure or blood pressure >140/90 millimeters of mercury (mmHg) at screening.
* Corrected QT interval (QTc) > 450 milliseconds.
* Where participation in study would result in donation of blood in excess of 500 mL within 56 days of starting the study.
* Subject whose calculated creatinine clearance is less than 80 mL/min
* Liver function tests above the upper limit of normal at screening (alkaline transaminase (ALT), aspartate transaminase (AST) or bilirubin).
* Chronic liver or biliary disease, history of Gilbert's syndrome in a previous clinical study or at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2007-09-05 (Actual); Primary Completion 2008-04-05 (Actual); Study Completion 2008-04-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal clinical chemistry findings | Up to 29 days
  Blood samples will be collected at specific time points as a measure of safety
Number of subjects with abnormal clinical hematology findings | Up to 29 days
  Blood samples will be collected at specific time points as a measure of safety
Number of subjects with abnormal urinalysis findings | Up to 29 days
  Urine samples will be collected at specific time points as a measure of safety
Number of subjects with abnormal blood pressure values | Up to 29 days
  Systolic and diastolic blood pressure will be measured in a supine position after at least 5 minutes of rest as a measure of safety.
Number of subjects with abnormal heart rate values | Up to 29 days
  Heart rate will be measured in a supine position after at least 5 minutes of rest as a measure of safety.
Number of subjects with abnormal respiratory rate values | Up to 29 days
  Respiratory rate will be measured in a supine position after at least 5 minutes of rest as a measure of safety.
Number of subjects with abnormal body temperature findings | Up to 29 days
  Body temperature will be measured in a supine position after at least 5 minutes of rest as a measure of safety.
Number of subjects with abnormal electrocardiogram (ECG) findings | Up to 29 days
  12-lead ECG measurements will be performed in a supine position after at least 5 minutes of rest as a measure of safety
Number of subjects with adverse events (AEs) | Up to 29 days
  An adverse event is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

SECONDARY OUTCOMES:
Plasma concentrations of GSK1827771 | Pre-dose, 0.25, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 1; in morning and evening on Day 2-7; in morning on Day 14, 21, 28
  Blood samples will be collected at specific time points for calculating plasma concentrations of GSK1827771
Maximum plasma concentration (Cmax) of GSK1827771 | Pre-dose, 0.25, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 1; in morning and evening on Day 2-7; in morning on Day 14, 21, 28
  Blood samples will be collected at specific time points for calculating Cmax of GSK1827771
Area under the curve (AUC) of GSK1827771 | Pre-dose, 0.25, 0.5, 1, 2, 4, 8, 12, 24 hours post-dose on Day 1; in morning and evening on Day 2-7; in morning on Day 14, 21, 28
  Blood samples will be collected at specific time points for calculating AUC of GSK1827771
Frequency of anti-GSK1827771 | Up to 29 days
  The presence of anti-GSK1827771 binding antibodies will be assessed using an immunoelectrochemiluminescence screening assay (ECL).
Titer of anti-GSK1827771 | Up to 29 days
  Blood samples for determination of anti-GSK1827771 antibodies will be taken at specific time points.
Frequency of anti-PEG | Up to 29 days
  Antibodies to PEG components of GSK1827771 will be measured.
Titer of anti-PEG | Up to 29 days
  Antibodies to PEG components of GSK1827771 will be measured.
Frequency of anti-dAb | Up to 29 days
  Antibodies to dAb components of GSK1827771 will be measured.
Titer of anti-dAb | Up to 29 days
  Antibodies to dAb components of GSK1827771 will be measured.
Change from Baseline response of whole blood to ex vivo stimulation with IL-1 alpha or IL-1 beta | Baseline and up to 29 days
  Blood samples will be collected for assessment of pharmacodynamic activity of GSK1827771 at specific time points
Exploratory biomarker levels in blood | Up to 29 days
  Blood samples will be taken for exploratory biomarker analysis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Baltimore, Maryland